CLINICAL TRIAL: NCT07207694
Title: The Effect of WhatsApp-Supported Education and Counseling on Healthy Lifestyle Behaviors, Glycemic Control, and Knowledge Levels in Patients With Stroke
Brief Title: WhatsApp-Based Education Program for Stroke Patients
Acronym: WEPS-P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nilgün Aras, Ph.D., Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-34215015-771; E-34215015 (Other: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital)
Record Dates: First submitted 2025-09-25; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Stroke
Keywords: Healthy Lifestyle Behaviors; type 2 diabetes mellitus; stroke
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Participants in the control group will receive routine face-to-face diabetes education and insulin injection training provided during hospitalization. The education is delivered verbally to patients and their caregivers by the clinical staff. After the follow-up period and data collection are completed, participants in the control group will also be offered access to the WhatsApp-based educational materials used in the intervention group.
  Interventions: Behavioral: Active Comparator: Routine Education
- WhatsApp-based education group (Experimental): Participants in the intervention group will receive the same routine face-to-face diabetes education and insulin injection training as the control group, plus a structured WhatsApp-based educational program. The WhatsApp intervention will be delivered over four weeks and include booklets/brochures, photos, and videos on diabetes definition and symptoms, complications, recognition and management of hypoglycemia and hyperglycemia, foot care, nutrition, exercise, oral antidiabetic and insulin therapy, and insulin injection demonstration. Participants' questions will be answered through WhatsApp to provide interactive support.
  Interventions: Behavioral: WhatsApp-based education group

INTERVENTIONS:
Behavioral: WhatsApp-based education group — Participants in the intervention group will receive the same routine face-to-face diabetes education and insulin injection training as the control group, plus a structured WhatsApp-based educational program. The WhatsApp intervention will be delivered over four weeks and include booklets/brochures, photos, and videos on diabetes definition and symptoms, complications, recognition and management of hypoglycemia and hyperglycemia, foot care, nutrition, exercise, oral antidiabetic and insulin therapy, and insulin injection demonstration. Participants' questions will be answered through WhatsApp to provide interactive support.
  Arms: WhatsApp-based education group
Behavioral: Active Comparator: Routine Education — Participants in the control group will receive routine face-to-face diabetes education and insulin injection training provided during hospitalization. The education is delivered verbally to patients and their caregivers by the clinical staff. After the follow-up period and data collection are completed, participants in the control group will also be offered access to the WhatsApp-based educational materials used in the intervention group.
  Arms: control group

SUMMARY:
Stroke is one of the leading causes of death and disability worldwide, with type 2 diabetes mellitus (T2DM) being a major risk factor that doubles the risk of ischemic stroke. Glycemic dysregulation is observed in nearly two-thirds of patients after acute stroke and is associated with both the severity of the initial cerebrovascular event and the risk of recurrence. Effective glycemic control, patient education, and adherence to treatment are therefore critical for secondary stroke prevention and improved patient outcomes.

Mobile health technologies, particularly social media applications, have become increasingly important in supporting chronic disease management. WhatsApp-based education has been shown to improve self-efficacy, self-management, and diabetes knowledge in patients with T2DM. However, there is a limited number of studies investigating the effect of WhatsApp-supported education and counseling on stroke patients with T2DM, especially regarding healthy lifestyle behaviors, glycemic control, and disease-related knowledge.

This randomized controlled trial aims to evaluate the effect of WhatsApp-supported education and counseling on healthy lifestyle behaviors, glycemic control, and knowledge levels among stroke patients receiving insulin therapy. Participants will be randomly assigned to either the intervention group or the control group. The control group will receive routine face-to-face diabetes education and insulin injection training during hospitalization. The intervention group will receive the same routine education plus a structured WhatsApp-based diabetes education program over four weeks. Educational content will include videos, photos, and booklets focusing on diabetes definition and symptoms, complications, hypoglycemia and hyperglycemia management, foot care, nutrition, exercise, oral antidiabetic and insulin therapy, and insulin injection demonstration. Participants' questions will be answered through WhatsApp messages, supporting continuous learning and adherence after discharge.

A total of 84 participants (42 per group) will be included, based on power analysis with a 5% significance level, 95% power, and accounting for a 10% dropout rate. Randomization will be conducted using block randomization with six combinations via an independent researcher through an online randomization tool. Data will be collected at baseline (T0) and six months after the intervention (T1). The primary outcomes include diabetes knowledge measured by the Revised Diabetes Knowledge Test-2, healthy lifestyle behaviors assessed using the Healthy Lifestyle Behavior Scale, and glycemic control parameters (fasting glucose, fasting insulin, HbA1c, and HOMA-IR).

All assessments will be performed by a trained nurse in the stroke clinic. Data analysis will include descriptive statistics, parametric or non-parametric tests depending on distribution, and reliability analyses using Cronbach's alpha. Ethical approval has been obtained from the Ethics Committee of SBÜ Gaziler Physical Training and Rehabilitation Research Hospital (Approval No: E-34215015).

This study is expected to demonstrate that WhatsApp-supported education and counseling improve patient knowledge, promote healthy lifestyle behaviors, and enhance glycemic control in stroke patients with T2DM. These findings may support the integration of digital counseling interventions into rehabilitation programs for secondary prevention and long-term disease management.

DETAILED DESCRIPTION:
Stroke remains the second leading cause of mortality and long-term disability worldwide. Type 2 diabetes mellitus (T2DM) is a well-established risk factor, doubling the risk of ischemic stroke compared with non-diabetic individuals. Glycemic dysregulation occurs in approximately two-thirds of patients after acute stroke and is directly correlated with both the severity of the acute cerebrovascular event and the likelihood of recurrence. Persistent poor glycemic control following stroke further increases the risk of recurrent events and reflects poor adherence to treatment regimens. Therefore, interventions that enhance glycemic control and promote adherence are of paramount importance in the secondary prevention of stroke among T2DM patients.

Educational and counseling interventions play a central role in diabetes self-management. Timely and appropriate insulin administration is essential for maintaining blood glucose levels within target ranges. Previous studies have demonstrated that structured diabetes and insulin education improves patients' glycemic outcomes and treatment adherence. In recent years, mobile health technologies and digital platforms have been increasingly used to support self-management and education. WhatsApp, a widely available and user-friendly communication platform, has proven effective in improving diabetes knowledge, self-efficacy, and self-management behaviors in individuals with T2DM. Nevertheless, there is a paucity of research evaluating the use of WhatsApp-based education and counseling specifically in stroke patients with coexisting T2DM, despite their high vulnerability to complications and recurrent stroke.

This randomized controlled trial was designed to address this gap by investigating the effectiveness of WhatsApp-supported education and counseling in improving healthy lifestyle behaviors, glycemic control, and knowledge levels among stroke patients undergoing insulin therapy. The study will be conducted at SBÜ Gaziler Physical Training and Rehabilitation Research Hospital.

Eligible participants will be adults aged 18 years and older with a diagnosis of ischemic stroke and T2DM, a Mini-Mental Test score greater than 18, and who are receiving insulin therapy. Exclusion criteria include incomplete data collection, major organ failure, or severe T2DM-related complications (e.g., diabetic foot, nephropathy, cardiovascular disease). Based on power analysis using a prior study on diabetes knowledge improvement, a total of 84 participants (42 in each group) will be recruited. Randomization will be performed in a 1:1 ratio using block randomization with four-unit blocks and six possible combinations, conducted independently via an online randomization tool (randomizer.org).

The control group will receive routine face-to-face diabetes education and insulin injection training delivered verbally during hospitalization. The intervention group will receive the same routine education plus a structured four-week WhatsApp-based education program. The WhatsApp intervention will deliver weekly educational content, including booklets, photos, and videos, covering the following topics:

Week 1: Definition, types, and symptoms of T2DM

Week 2: Complications of T2DM; recognition and management of hypoglycemia and hyperglycemia; importance of foot care

Week 3: Nutrition and exercise in diabetes management

Week 4: Diabetes treatment, including oral antidiabetic agents, insulin therapy, and insulin injection demonstration

In addition, participants in the intervention group will be able to ask questions through WhatsApp, which will be answered by the research team to ensure interactive and continuous support.

Data will be collected at baseline (T0) and six months after the intervention (T1). Tools include the Revised Diabetes Knowledge Test-2 (23 items), the Healthy Lifestyle Behavior Scale (34 items, 5-point Likert), and a demographic/clinical data form including sociodemographic characteristics, comorbidities, medications, fasting glucose, fasting insulin, HbA1c, and HOMA-IR levels. The Revised Diabetes Knowledge Test-2 has been validated in Turkish, and the Healthy Lifestyle Behavior Scale has demonstrated high reliability (Cronbach's alpha = 0.86).

All assessments will be conducted by a trained nurse in the stroke clinic. Data analysis will use SPSS software, applying descriptive statistics, normality tests, and appropriate parametric or non-parametric tests. Reliability will be assessed using Cronbach's alpha. A p-value of <0.05 will be considered statistically significant.

Ethical approval has been granted by the Ethics Committee of SBÜ Gaziler Physical Training and Rehabilitation Research Hospital (Approval No: E-34215015). Written informed consent will be obtained from all participants prior to enrollment.

The study is expected to demonstrate that WhatsApp-supported education and counseling, when integrated with routine hospital-based education, enhance patient knowledge, foster healthier lifestyle behaviors, and improve glycemic control in stroke patients with T2DM. If proven effective, this intervention may provide an accessible, cost-effective, and scalable approach for integrating mobile health tools into rehabilitation nursing and chronic disease management programs, ultimately contributing to better long-term outcomes and reduced recurrence of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of ischemic stroke
* Mini-Mental Test (MMT) score > 18
* Receiving insulin therapy for type 2 diabetes mellitus (T2DM)
* Ability to use WhatsApp on a smartphone (participant or caregiver)
* Willingness to provide informed consent

Exclusion Criteria:

* Presence of major organ failure
* Development of severe T2DM-related complications (e.g., diabetic foot, nephropathy, cardiovascular disease)
* Cognitive or communication impairments preventing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Diabetes Knowledge | Baseline (T0) and 6 months after intervention (T1)
  Assessed using the Revised Diabetes Knowledge Test-2 (23 items). Scores range from 0 to 23, with higher scores indicating greater diabetes knowledge.
Change in HbA1c | Baseline (T0) and 6 months after intervention (T1)
  Laboratory value HbA1c (%). Lower levels indicate better glycemic control.
Change in Healthy Lifestyle Behaviors | Baseline (T0) and 6 months after intervention (T1)
  Measured by the Healthy Lifestyle Behavior Scale (34 items, 5-point Likert). Scores range from 0-100, with higher scores reflecting healthier lifestyle behaviors
Change in fasting glucose | Baseline (T0) and 6 months after intervention (T1)
  Laboratory value: fasting glucose (mg/dL). Measurement of blood glucose levels after at least 8 hours of fasting. Lower values indicate better glycemic control.
Change in fasting insulin | Baseline (T0) and 6 months after intervention (T1)
  Laboratory value: fasting insulin (µIU/mL). Measurement of circulating insulin levels after at least 8 hours of fasting. Lower levels indicate improved insulin sensitivity and better glycemic control.
Change in HOMA-IR | Baseline (T0) and 6 months after intervention (T1)
  Laboratory value: HOMA-IR (Homeostatic Model Assessment of Insulin Resistance). Calculated from fasting glucose and fasting insulin using the formula:
  HOMA-IR=Fasting Glucose (mg/dL)×Fasting Insulin (µIU/mL):405
  Higher values indicate greater insulin resistance, whereas lower values reflect better glycemic control.

IPD SHARING:
Plan to Share IPD: No